CLINICAL TRIAL: NCT00666393
Title: An Open-Label Evaluation of Safety of the IONSYS System [Fentanyl Iontophoretic Transdermal System (40ug) for Management of Acute Post-Operative Pain in Pediatric Patients
Brief Title: An Evaluation of Safety of the Fentanyl Transdermal System for Management of Acute Post-Operative Pain in Pediatric Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Program Cancelled.
Sponsor: Alza Corporation, DE, USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013048; C-2006-007 (Other: Alza Corporation, DE, USA)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Pain, Postoperative; Pediatrics
Keywords: IONSYS™; Pain, Postoperative; Analgesia, Patient-Controlled; Opioids; Pediatrics
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental)
  Interventions: Drug: fentanyl iontophoretic transdermal system (40mcg) No placebo; Drug: fentanyl iontophoretic transdermal system (40mcg)

INTERVENTIONS:
Drug: fentanyl iontophoretic transdermal system (40mcg) No placebo — 40 mcg per dose, maximum of 6 doses/hour; total maximum 80 doses/24 hours
Drug: fentanyl iontophoretic transdermal system (40mcg) — 40 mcg per dose, maximum of 6 doses/hour; total maximum 80 doses/24 hours

SUMMARY:
The purpose of this study is to evaluate the safety and clinical utility of fentanyl HCl 40 mcg system for the management of postoperative pain in pediatric inpatients.

DETAILED DESCRIPTION:
This will be a multicenter, open-label study in which hospitalized pediatric post-operative patients will receive the fentanyl HCl 40 mcg system for up to 3 consecutive days. After their surgery, patients will be brought to the recovery room for initial observation following general or regional anesthesia for abdominal, pelvic/genitourinary, orthopedic, or thoracic surgery. Post surgery procedures will be preformed and when analgesia is required, the patient will be titrated to analgesic comfort (a pain score < 4 on a scale 0-10) for at least 30 minutes with an intravenous opioid as clinically appropriate. After a patient has been comfortable (pain intensity of < 4 on 0 -10 color visual analog scale ) for > 30 minutes and has been monitored during recovery and is awake, able to answer questions and follow commands he/she will be assessed for pain intensity, vital signs, and oxygen saturation (amount of oxygen in the blood). If the patient meets study entry criteria, baseline assessments (pain intensity, vital signs, and oxygen saturation) will be completed and the fentanyl HCl 40 mcg system will be applied. During the first 3-hours of the treatment, if a patient successfully completed an on-demand dose and pain relief was still inadequate, the patient could deliver another dose of fentanyl, or be re-titrated to comfort with single or multiple intravenous doses of supplemental opioid medication (IV fentanyl or IV morphine) per study physician's clinical discretion. Supplemental IV doses of opioid medications can be administered in the first 3-hours of system application, but are prohibited after Hour 3. If pain control is judged inadequate with the combined use of fentanyl HCl 40 mcg system and the use of supplemental analgesia, the patient may be withdrawn from the study. Patients will receive fentanyl HCl 40 mcg system. Fentanyl will be delivered upon patient activation over 10 minutes for a maximum of 6 doses/hour for up to 24 hrs or 80 total doses whichever occurs first for up to three consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* The patients must: weigh >= 40 kg
* be scheduled for abdominal, pelvic/genitourinary, orthopedic, or thoracic surgery
* Be expected by the investigator's staff to require injected opioid analgesia for at least 24 hours after surgery
* Be judged by the investigator's staff to be capable of understanding and cooperating with the requirements of the study.

Exclusion Criteria:

* Patients who have undergone any surgery on the airway, head or neck
* Patients who are expected to require intensive care
* Patients who require airway(breathing) support after their surgery
* Patients who received intra-operative (during surgery) and/or post-operative (after surgery) administration of opioids other than morphine, hydromorphone, fentanyl, sufentanil or alfentanil
* Patients with active generalized skin disorders or active local skin disease that precludes the application of fentanyl iontophoretic transdermal system(40 mcg).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Any adverse events will be recorded. Oxygen saturation will be monitored continuously. Vital signs (BP, HR, RR, T), oxygen saturation, and concomitant medications will be recorded at Hours 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and every 4 hours thereafter. | Safety outcomes will be collected at intervals throughout the drug system application for a maximum of 72 hours.

SECONDARY OUTCOMES:
Patient Global Assessment, Investigator Global Assessment and Parent Assessment of Patient Use will be completed every 24 hours. Serum fentanyl concentration will be collected at Hours 3, 6,12, and 24. | Patient, Investigator and Parent Assessments of the treatment will be completed every 24 hours for a maximum of 72 hours. Pharmacokinetic measurements will be completed 4 times during every 24 hours of treatment for a maximum of 12 times over 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA